CLINICAL TRIAL: NCT06106607
Title: Physical Activity and Sedentary Behaviour in Patients With Inflammatory Bowel Disease - Epidemiology and Interventions
Brief Title: Physical Activity and Sedentary Behaviour in Patients With Inflammatory Bowel Disease
Acronym: PASIBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Clinical Research and Prevention (Network)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Tanja Thomsen, Postdoc, Center for Clinical Research and Prevention
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-22040390
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Inflammatory Bowel Diseases; Physical Activity; Sedentary Behavior; Feasibility Study
MeSH Terms: conditions — Inflammatory Bowel Diseases; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Allocation status of study participants will not be revealed for the project nurses that conduct the outcome assessments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This group will undergo a 20-week individually tailored, behavioral intervention
  Interventions: Behavioral: Intervention group
- Control group (No Intervention): This group will be encouraged to maintain usual lifestyle and activities.

INTERVENTIONS:
Behavioral: Intervention group — A 20-week intervention with a basic part, including
  1. A group session with education about IBD,physical activity and exercise in relation to IBD (definitions, evidence and recommendations). Furthermore, access to a video with general information about IBD, physical activity and exercise
  2. Four individual motivational counselling sessions (two physical, two by telephone) with a project nurse. These will involve identifying individual motivation and opportunities for increasing physical activity and behavioral goal setting.
  An optional intervention part will follow, including choises between (or all of)
  1. A one-hour individual session with a physiotherapist, involving guidance in physical activity and exercise tailored to the individual.
  2. Being teamed up with 1-2 'exercise buddies' (other participants from the overall intervention group).
  3. Access to 4 short 2-3 minutes videos/'reels' of a physiotherapist explaining and demonstrating beneficial physical exercises.
  Arms: Intervention group

SUMMARY:
Emerging research suggests that physical activity may improve health-related quality of life (HrQoL) in patients with inflammatory bowel disease (IBD) and positively influence physical symptoms, fatigue, stress and anxiety. However, little is known about detailed movement patterns and their specific health effects in IBD patients or about patients' wishes, motivation and preferences for physical activity in their everyday lives.

Based on exisiting evidence, the investigators' hypothesis is that an individually tailored, behavioural intervention focusing on reducing sedentary behaviour and increasing daily physical activity is feasible and effective in patients with IBD. Therefore, the overall aim of this randomized feasibility study is to determine the feasibility of the behavioural intervention, including the testing of recruitment procedures, intervention adherence, retention and outcome assessments.

Intervention participants will undergo:

1. A group session with information about IBD and the effects and recommendations of physical activity and exercise
2. Four motivational interviews with a project nurse, including goal-setting and action plans
3. An optional part, where each participant will have the possibility of choosing between:

   * An one-hour individual session with a physiotherapist
   * Being teamed up with 1-2 'exercise buddies' (other intervention participants) and/or
   * Access to four short 2-3 minutes videos/'reels' of a physiotherapist explaining and demonstrating beneficial physical exercises

Results from the present feasibility study will determine if and how to proceed with a large-scale randomized controlled trial evaluating the efficacy of the intervention.

DETAILED DESCRIPTION:
Although existing literature indicates potential health benefits of physical activity and exercise in patients with IBD, there is little consistency in the proposed interventions for promoting physical activity, and large variations in the applied physical activity intensities and types in the existing physical activity intervention studies. Patients with IBD experience barriers to engaging in physical activity that are related to both stigmatization and disease symptoms. These are barriers that might be overcome if the physical intervention is focusing on variation in physical activity intensity and is tailored to the individual patient. The investigators' hypothesis is that an individually tailored, behavioural intervention focusing on physical activity in a 24-hour perspective, including sedentary behaviour and physical activity from light to vigorous intensity, is feasible and effective in patients with IBD.

The present feasibility study aims to test the behavioural intervention for feasibility and acceptability in a small sample (N=30) of patients with IBD from the gastroenterology outpatient clinic at Bispebjerg Hospital, Copenhagen, Denmark. By conducting a feasibility study with a small sample size, the investigators want to follow the course and applicability of an intervention that has been developed as an individual offer with possibilities and solutions for the individual patient, but still operated within a controlled and standardized research frame. Assessment of feasibility will include identification of barriers for recruitment, acceptance of group/randomization status, delivery methods, retention, outcome assessments and logistics. Outcome measures that will be tested for feasibility include objectively measured physical activity levels (over a 7-day period), health-related quality of life, fatigue, pain, mental health and cardio-metabolic biomarkers.

The intervention will address the individual patient's knowledge, motivation, resources and opportunities for reducing sedentary behaviour and increasing daily physical activity and exercise in the individual's everyday life.

The 20-week intervention will consist of a basic part for all participants, which will include

1. A group session with education about IBD in general and about physical activity and exercise in relation to IBD (definitions, evidence and recommendations). Following this session, the participants will also be offered access to a video with general information about IBD, physical activity and exercise
2. Four individual motivational counselling sessions (two physical and two telephone sessions) with a project nurse. The counselling sessions will involve identifying the individual's motivation and opportunities for increasing physical activity, behavioral goal setting and action planning.

An optional intervention part will then follow, where the individual participant will have the possibility of choosing between (or all of)

1. A one-hour individual session with a physiotherapist from Bispebjerg/Frederiksberg Hospitals, which will involve guidance in physical activity and exercise tailored to the individual participant. This could be the case if a participant experiences specific symptoms or limitations when engaging in physical activity and/or exercise and needs individual guidance related to this.
2. Being teamed up with 1-2 'exercise buddies' (other participants from the overall intervention group).
3. Access to 4 short 2-3 minutes videos/'reels' of a physiotherapist explaining and demonstrating beneficial physical exercises. The videos aim to provide participants with new inspiration and practical suggestions to increase their physical activity and exercise.

The main setting of the intervention will be the participants' everyday lives (family, work/school, leisure-time activities). However, the Gastroenterology Department, Bispebjerg Hospital, and potentially, local municipal health centres and sports clubs will be the actual physical places for the specific intervention elements (e.g. education, counselling sessions, physiotherapist-led sessions, exercising in small communities ('exercise buddies').

Participants randomized to the control group will be encouraged to maintain their usual lifestyle and activities. They will be expected to undergo the same baseline - and outcome assessment as the participants in the intervention group.

Results from the present feasibility study will determine if and how to proceed with a large-scale randomized controlled trial evaluating the efficacy of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of IBD (Crohn's disease or ulcerative colitis) > 1 year
* Over 18 years of age
* Minimum three months stable medication type and dose without use of steroids as part of the medical treatment during the last three months
* Speak and understand Danish

Exclusion Criteria:

* Unable to give informed consent
* Active inflammatory disease in joints, skin, pancreas, thyroid, lungs or liver that can hinder engagement in physical activity and exercise
* Cognitive and/or mental disabilities that can hinder engagement in physical activity and exercise
* Engaging in high-intensity physical activity -/> 8 hours pr week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
Recruitment | Assessed at 3 months after baseline
  Recruitment rates will be calculated as the proportion of patients randomised/proportion of patients eligible
Retention | Assessed at 5 months (20 weeks)
  Retention rates will be calculated as the proportion of patients providing the outcomes of interest/proportion of patients randomised
Intervention adherence | Assessed at 5 months (20 weeks)
  Adherence to intervention protocol will be calculated as the number of group and motivational counselling sessions attended out of the total number of sessions available
Intervention acceptability | Assessed at 5 months (20 weeks)
  Acceptability of intervention protocol will be calculated as the number of received optional elements of the intervention out of the total number of optional intervention elements available

SECONDARY OUTCOMES:
Objectively measured physical activity measured by SENS monitor | Assessed at baseline and at 5 months (20 weeks)
  The SENS Motion sensor is an activity sensor, which captures seven-day, 24-hour physical activity patterns, including number of steps and the amount of daily time lying down, sitting, standing, and being active with light, moderate and high intensity, as well as specific activities such as bicycling or walking stairs
Self-reported physical activity and sitting time measured by the Physical Activity Scale (PAS) | Assessed at baseline and at 5 months (20 weeks)
  Self-reported physical activity (light, moderate, vigorous) and sitting time at work and during leisure time will be measured by the Physical Activity Scale 2.1 (PAS 2.1). Participants will be asked to specify number of hours and minutes in an average 24-hour day spent sitting at work and during leisure time. In addition, participants will report number of weekly hours and minutes spent in light, moderate or vigorous intensity activities.
Exercise self-efficacy measured by the Exercise Self-Efficacy Scale | Assessed at baseline and at 5 months (20 weeks)
  The Exercise Self-Efficacy Scale assesses an individual's beliefs in their ability to continue exercising under different circumstances.
Health-related quality of life measured by the Inflammatory Bowel Disease Questionnaire (IBDQ) | Assessed at baseline and at 5 months (20 weeks)
  Quality of life will be measured by the 32-item Inflammatory Bowel Disease Questionnaire (IBDQ-32). The IBDQ-32 captures the patient's experience of IBD on four domains of functioning and well-being: 1) bowel symptoms, 2) systemic symptoms, 3) emotional function and 4) social function.
Fatigue measured by The Multi-dimensional Fatigue Inventory (MFI-20) | Assessed at baseline and at 5 months (20 weeks)
  Fatigue will be measured by the 20-item Multi-dimensional Fatigue Inventory (MFI 20) . MFI 20 consists of 20 statements, which classifies fatigue in five dimensions: 1) general fatigue 2) physical fatigue 3) mental fatigue 4) reduced activity 5) reduced motivation.
Fatigue measured by the visual analogue scale for fatigue (VAS-Fatigue) | Assessed at baseline and at 5 months (20 weeks)
  Fatigue measured by the visual analogue scale for fatigue (VAS-fatigue). Score from 0-100. Higher score is more fatigue.
Pain intensity measured by the visual analogue scale for pain (VAS-Pain) | Assessed at baseline and at 5 months (20 weeks)
  Pain will be measured by the visual analogue scale for pain. Score from 0-100. The higher score, the higher pain intensity.
Mental health measured by The Hospital Anxiety and Depression Scale (HADS) questionnaire | Assessed at baseline and at 5 months (20 weeks)
  The HADS questionnaire consists of seven items for depression and anxiety subscales, respectively. Scoring for each item ranges from zero to three, with three indicating highest anxiety or depression level.
IBD-related disease activity measured by fecal calprotectin | Assessed at baseline and at 5 months (20 weeks)
  Fecal calprotectin is a stool test that is used to detect inflammation in the intestines. It will be used to monitor the participants' disease activity and severity.
Serum lipids measured by blood sample | Assessed at baseline and at 5 months (20 weeks)
  Total cholesterol, high-density lipoprotein cholesterol (HDL), and triglycerides will be measured by a blood sample. Low-density lipoprotein cholesterol (LDL) will be calculated.
Glycosylated hemoglobin (HbA1c) measured by blood sample | Assessed at baseline and at 5 months (20 weeks)
  Glycosylated hemoglobin, type A1c (HbA1c) will be determined by a blood sample
Disease activity measured by a C-Reactive Protein (CRP) test | Assessed at baseline and at 5 months (20 weeks)
  A venous blood sample will be drawn (not fasting)
Blood pressure measurements | Assessed at baseline and at 5 months (20 weeks)
  Blood pressure will be measured, after 5 to 10 minutes of rest, 3 times at the right upper arm (average of the 3 measurements) with the participant in a sitting/lying position.
Body weight in kilograms | Assessed at baseline and at 5 months (20 weeks)
  Body weight is measured in light clothing without shoes to the nearest 0.1 kg
Waist circumference measured in centimeters | Assessed at baseline and at 5 months (20 weeks)
  Waist circumference will be measured midway between the lower rib margin and the iliac crest to the nearest 0.5 centimeter, without any pressure to the skin and with an unstretched tape measure.
Hip circumference measured in centimeters | Assessed at baseline and at 5 months (20 weeks)
  Hip circumference will be measured at the point yielding the maximum circumference over the buttocks to the nearest 0.5 centimeter. The tape measure will be be held in a horizontal plane touching the skin but not indenting the soft tissue.
Waist-hip-ratio | Assessed at baseline and at 5 months (20 weeks)
  Waist-hip-ratio will be calculated based on the assessments of waist and hip circumferences
Body mass Index (BMI) | Assessed at baseline and at 5 months (20 weeks)
  Body mass Index (BMI, kg/m2) will be calculated based on the assessment of body weight and height.

CONTACTS AND LOCATIONS:
Overall Officials: Mette Aadahl, PhD, Principal Investigator — Professor at Center for Clinical Research and Prevention
Locations (1):
- Digestive Disease Center, BFH, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
As this is a feasibility study, sharing of outcome data is not relevant

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT06106607/Prot_SAP_000.pdf